CLINICAL TRIAL: NCT01752816
Title: Does Aerobic Training Followed by Resistance Training Enhance Aerobic Capacity in Seniors? A Randomized Controlled Trial.
Brief Title: Does Aerobic Training Followed by Resistance Training Enhance Aerobic Capacity in Seniors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Gisela Sjogaard, professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S-20120178
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-04

CONDITIONS: Elderly
Keywords: endurance training,; strength training,; aerobic capacity,; muscle strenght; physical capacity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endurance training (Active Comparator): 40 min bicycle or treadmill training at 60% maximal oxygen uptake
  Interventions: Behavioral: exercise training
- Strength following endurance training (Experimental): 20 minutes bicycle or treadmill training at 60% maximal oxygen uptake followed by 20 minutes stength training increasing from 15RM to 10RM
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training

SUMMARY:
In healthy young subjects a single bout of strength training following endurance training has been shown to improve markers for aerobic capacity in muscle compared to a single bout of endurance training alone. The present project tests the hypothesis: 12 weeks of training with sessions of endurance training followed by strength training is superior to endurance training alone for health participants 50-65 years of age. The outcome measures are maximal oxygen uptake and knee-extension strength.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* understanding Danish language

Exclusion Criteria:

* medical contraindication for training
* taking beta-blockers
* physical exercise training more than 2 hrs per week

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
maximal oxygen uptake | 12 weeks
knee extension strength | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Sjøgaard, DrMedSci, Principal Investigator — University of Southern Denmark
Locations (1):
- Næstved Senior Motion klub, Næstved, Region Sjælland, Denmark

REFERENCES:
- See also: Research Unit: Physical Activity and Health at Work — http://www.sdu.dk/en/Om_SDU/Institutter_centre/Iob_Idraet_og_biomekanik/Forskning/Forskningsenheder/FysiskAktivitetSundhed